CLINICAL TRIAL: NCT05096234
Title: Pilot Study of [18F]F-AraG PET Imaging to Evaluate Immunological Response to Chimeric Antigen Receptor (CAR) T Cell Therapy in Lymphoma
Brief Title: 18F-F-AraG PET Imaging to Evaluate Immunological Response to CAR T Cell Therapy in Lymphoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: loss of sponsor support
Sponsor: Stanford University (Other)
Collaborators: CellSight Technologies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB-56655; CCT5038 (Other: OnCore)
Record Dates: First submitted 2021-10-14; First posted 2021-10-27 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- [18F]F-AraG PET (Experimental): Subjects will undergo PET imaging at the following time points:
  * Baseline, prior to lymphodepleting chemotherapy: [18F]F-AraGPET/CT, followed the next day by FDG-PET/CT
  * At peak CAR expansion: Day 4 (± 2 days) post-CAR infusion:
    [18F]F-AraG PET
  * At Day +28 (± 4 days) post-CAR infusion: FDG-PET/CT Subjects will have a paired biopsy after each imaging time point, if possible. Subjects will be followed for safety of [18F]F-AraG for 30 days after last dose
  Interventions: Drug: [ 18F]F-AraG PET

INTERVENTIONS:
Drug: [ 18F]F-AraG PET — Dose: 5 mCi (±10%) Mode of Administration: Intravenous (IV)
  Other Names: [ 18F]F-AraG (2'-deoxy-2'-fluoro-9-β-D- arabinofuranosylguanine; trade name VisAcT)

SUMMARY:
This is a pilot study in adult subjects with aggressive B-cell lymphoma who will receive commercial or research CAR T cell therapy as anticancer treatment.

DETAILED DESCRIPTION:
Primary Objectives:

* Explore the relationship of change in [18F]F-AraG PET signal following CAR T cell treatment with changes in T cell infiltration in tumor biopsies.

Exploratory Analyses:

* Explore the relationship of change in [18F]F-AraG PET signal in tumor lesions following CAR T cell treatment with clinical benefit rate (defined as Complete Response (CR) + Partial Response (PR) + stable disease (SD) ≥ 3 months) using RECISTv1.1 criteria
* Correlate the change in [18F]F-AraG PET signal in tumor lesions following CAR T cell therapy with maximum grade of Cytokine Release Syndrome (CRS) and neurotoxicity experienced.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Histologically confirmed aggressive B cell NHL including the following types defined by WHO 2008:

  * DLBCL not otherwise specified; T cell/histiocyte rich large B cell lymphoma; DLBCL associated with chronic inflammation; Epstein Barr virus (EBV)+ DLBCL of the elderly; OR
  * primary mediastinal (thymic) large B cell lymphoma
  * transformation of follicular lymphoma, marginal zone lymphoma or chronic lymphocytic leukemia to DLBCL will also be included
* Measurable disease by PET imaging (as defined by Cheson (2014)), that meets all the following criteria:

  * At least one measureable lesion away from head & neck, liver, kidneys, GI tract and bladder
  * At least one biopsy-accessible lesion or lymph node.
* Express willingness to undergo low risk FNA or core biopsy of subcutaneous accessible lesion or lymph node.
* Scheduled to receive commercial or research CAR T cell therapy with axicabtagene ciloleucel (Yescarta ®) as part of anticancer therapy.
* Adequate renal and hepatic function, defined as:

  1. Creatinine clearance (as estimated by Cockcroft Gault) ≥ 60 mL/min or Cr < 1.6 mg/dL
  2. Serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≤ 2.5x upper limit of normal (ULN)
  3. Total bilirubin ≤ 1.5 mg/dL, except in cases of Gilbert's syndrome
* Able to give informed consent. Subjects unable to give informed consent will not be eligible for this study

Exclusion Criteria:

* Women who are pregnant or breastfeeding.
* Subjects with significant GI disease involvement by PET imaging
* In the investigator's judgment, have any medical condition likely to interfere with assessment of safety or efficacy, be unable to tolerate additional radiation, or be unlikely to complete all protocol-required visits and procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2021-09-28 (Actual); Primary Completion 2022-05-09 (Actual); Study Completion 2023-10-09 (Actual)

PRIMARY OUTCOMES:
Primary outcome measure | values obtained on Day 0 and Day 4 (± 2 days)
  Spearman correlation between changes in SUV in [18F]F-AraG signal on PET imaging to changes in T-cell infiltrates in biopsy samples

OTHER OUTCOMES:
First exploratory outcome measure | ≥ 3 months
  correlation between changes in SUV [18F]F-AraG signal on PET imaging to the observed clinical benefit rate using RECISTv1.1 criteria.
Second exploratory outcome measure | ≥ 3 months
  Correlation between changes in [18F]F-AraG signal to the frequency and grade of two common CAR T cell toxicities, cytokine release syndrome (CRS) and neurotoxicity, if observed in this study population.

CONTACTS AND LOCATIONS:
Overall Officials: David Miklos, MD, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No